CLINICAL TRIAL: NCT00977314
Title: Bone Conduction Auditory Performance Via the Tooth for Single-Sided Deafness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonitus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN002
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Unilateral Hearing Loss
Keywords: Unilateral Hearing Loss
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SoundBite Hearing System (Experimental): The objective of this study was to assess the safety and effectiveness of the SoundBite hearing system by Sonitus Medical and to support its intended use for the treatment of unilateral hearing loss. The SoundBite hearing system is a Bone Conduction Device (BCD) and is occasionally referred to as such in the protocol and within this report.
  Interventions: Device: The Sonitus Bone Conduction Hearing System; Device: SoundBite; Device: SoundBite Hearing System

INTERVENTIONS:
Device: The Sonitus Bone Conduction Hearing System — Comparison of HINT scores (Speech front with noise at better ear) at 30 days tested with the device in place verses with the device removed.
Device: SoundBite
Device: SoundBite Hearing System

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using bone conduction via the teeth to treat Single-Sided Deafness (SSD).

DETAILED DESCRIPTION:
The Sonitus Bone Conduction Device (BCD) is a bone conduction device for single-sided deafness (SSD). The Sonitus BCD consists of an Oral Appliance (OA), an external microphone component, worn behind the ear (BTE), a calibration interface cable and a PC-controlled calibration software for subject calibration. The Sonitus BCD picks up sounds from a microphone located within the ear canal of the deaf ear, capitalizing on the acoustics of the natural pinna and ear canal. The signal picked up by the microphone is then transmitted wirelessly to a removeable bone conduction oral appliance located on the upper molars. The oral appliance receives the acoustic signal from the BTE and applies an equivalent vibratory signal to the teeth that reaches the skull via bone conduction and routed transcranially to the contralateral cochlea.

ELIGIBILITY:
Inclusion Criteria:

* Must be >18, < 80 years old
* Must be fluent in English, as determined by the PI
* Must not be a member of a vulnerable group (IRB defined)
* Must remain in geographic area during duration of the study
* Diagnosis of acquired SSD (Section 3.1), time since onset (≥3 mos)
* Must have a minimum of 6 posterior teeth remaining in the upper arch (3 teeth per side),third molars are acceptable if healthy, fully erupted and substituting for second molars

Exclusion Criteria:

* Must not be current users of devices such as Baha, CROS or TransEar
* Must not have known active medical causes of SSD:

  * Active middle ear pathology
  * Conductive HL (Otosclerosis, otitis media, otitis externa and others)
  * Sudden hearing loss that is not stable
* Must not have known medical problems that might be life-threatening or is a contraindication for elective dental or medical procedures
* Must not have known problems that may interfere with the impression procedure, such as inability to breath through nose (e.g. severe flu, allergies or cold)
* Must not have allergies to polymers
* Must not have known dental abnormalities:

  * Temporary crowns or undergoing dental treatment
  * Poor oral hygiene and/or rampant decay
  * Current orthodontics
  * Active caries in one or more of the possible abutment teeth for the device
  * Active moderate to severe periodontal disease around abutment teeth for the device
  * Suspicious oral/facial lesions or swelling of any type
  * Severe pain on palpation on any area of mouth, face or neck
  * Moderate to severe heat sensitivity on any of the upper teeth
  * Subject currently being treated for temporomandibular joint disorder (TMJ), pain, full mouth reconstruction or posterior dental implants
* Must not have known Audiological conditions:

  * Conductive hearing loss (air-bone gap >10dB HL at more than 3 frequencies)
  * Word recognition scores inconsistent with pure tone averages
  * Fluctuating hearing loss
* Must not have known psychological factors that interfere with their ability to comply, comprehend, consent and cooperate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Murray, MD, Principal Investigator
Locations (2):
- United States (2):
  - Hearing Resource Center, Redwood City, California
  - Camino Ear Nose and Throat, San Jose, California

REFERENCES:
- [Background] Ozer E, Adelman C, Freeman S, Sohmer H. Bone conduction hearing on the teeth of the lower jaw. J Basic Clin Physiol Pharmacol. 2002;13(2):89-96. doi: 10.1515/jbcpp.2002.13.2.89. PMID 16411423
- [Background] Soli SD, Wong LL. Assessment of speech intelligibility in noise with the Hearing in Noise Test. Int J Audiol. 2008 Jun;47(6):356-61. doi: 10.1080/14992020801895136. No abstract available. PMID 18569108
- [Background] Dahlin GC, Allen FG, Collard EW. Bone-conduction thresholds of human teeth. J Acoust Soc Am. 1973 May;53(5):1434-7. doi: 10.1121/1.1913490. No abstract available. PMID 4712563
- [Background] Wazen JJ, Spitzer J, Ghossaini SN, Kacker A, Zschommler A. Results of the bone-anchored hearing aid in unilateral hearing loss. Laryngoscope. 2001 Jun;111(6):955-8. doi: 10.1097/00005537-200106000-00005. PMID 11404603
- [Background] Wazen JJ, Spitzer JB, Ghossaini SN, Fayad JN, Niparko JK, Cox K, Brackmann DE, Soli SD. Transcranial contralateral cochlear stimulation in unilateral deafness. Otolaryngol Head Neck Surg. 2003 Sep;129(3):248-54. doi: 10.1016/S0194-5998(03)00527-8. PMID 12958575
- [Background] Stenfelt SP, Hakansson BE. Sensitivity to bone-conducted sound: excitation of the mastoid vs the teeth. Scand Audiol. 1999;28(3):190-8. doi: 10.1080/010503999424761. PMID 10489868
- [Background] Murray M, Miller R, Hujoel P, Popelka GR. Long-term safety and benefit of a new intraoral device for single-sided deafness. Otol Neurotol. 2011 Oct;32(8):1262-9. doi: 10.1097/MAO.0b013e31822a1cac. PMID 21799455
- [Background] Miller R, Hujoel P, Murray M, Popelka GR. Safety of an intra-oral hearing device utilizing a split-mouth research design. J Clin Dent. 2011;22(5):159-62. PMID 22403981
- [Background] Popelka GR, Derebery J, Blevins NH, Murray M, Moore BC, Sweetow RW, Wu B, Katsis M. Preliminary evaluation of a novel bone-conduction device for single-sided deafness. Otol Neurotol. 2010 Apr;31(3):492-7. doi: 10.1097/MAO.0b013e3181be6741. PMID 19816229
- [Result] Murray M, Popelka GR, Miller R. Efficacy and safety of an in-the-mouth bone conduction device for single-sided deafness. Otol Neurotol. 2011 Apr;32(3):437-43. doi: 10.1097/MAO.0b013e3182096b1d. PMID 21221045
- See also: SoundBite Hearing Device — http://www.soundbitehearing.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment/Enrollment Phase(September 2009-November 2009) Location: Medical Clinics Meant to assess the subjects' ability to be enrolled in the trial, included Medical, Audiological and Dental evaluations.
Pre-assignment Details: Phase 1: Enrollment: Assesses the subjects' ability to be enrolled in the trial. It included medical, audiological, and dental evaluations and device fit to ensure comfort during the duration of the trial.
Groups:
- Analyzed Group: 30 subjects were enrolled in the analyzed group with only 24 subjects expected to complete it. With an approximated 20% subject dropout rate anticipated. The total number of subjects that completed the study was 28 of 30 enrolled in the analyzed group.
- Pilot Group: Per the protocol, the first five (5) subjects were enrolled in the "pilot group" of the study to work out the process flow and training of the centers and participants.
Period: Overall Study
Arm/Group | Analyzed Group | Pilot Group
Started | 30 | 5 (First 5 subjects enrolled were pilot subjects and not included in analysis.)
Completed | 28 | 5 (First 5 subjects enrolled were pilot subjects and not included in analysis.)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: 35 subjects were enrolled in this study.Per protocol,the first 5 subjects enrolled were the pilot phase of the study. Data obtained from the first 5 subjects were excluded from analyses.An approximated 20% subject dropout rate anticipated, 30 subjects were enrolled with 24 subjects expected complete.
Groups:
- Analyzed Group; Pilot Group: A total of thirty-five (35) subjects were enrolled in this study. Per the protocol, the first five (5) subjects enrolled were the pilot phase of the study to work out the process flow and training of the centers and participants. The data obtained from the first five subjects were excluded from all analyses. With an approximated 20% subject dropout rate anticipated, 30 subjects were enrolled in the study with only 24 subjects expected to complete it.
- Total: Total of all reporting groups
Arm/Group | Analyzed Group | Pilot Group | Total
Number analyzed (Participants) | 30 | 5 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 5 | 34
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (13) | 45.4 (8.1) | 46.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 18
  Male | 15 | 2 | 17
Region of Enrollment [Number; unit: participants]
  United States | 30 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Device- and Procedure-related Adverse Events at 30 Days
Description: The safety parameters for the trial were monitored throughout the Evaluation Phase (30 days). The safety checks included:
  Comprehensive Medical evaluation at Enrollment and at Termination Comprehensive Dental evaluation at Enrollment and at Termination, with interim dental checks at each visit in between, if needed Comprehensive Audiological evaluation at Enrollment and Termination.
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Medical, Dental, Audiological Safety 30 Days: The safety parameters for the trial were monitored throughout the Evaluation Phase (30 days). The safety checks included:
  * Comprehensive Medical evaluation at Enrollment and at Termination
  * Comprehensive Dental evaluation at Enrollment and at Termination, with interim dental checks at each visit in between, if needed
  * Comprehensive Audiological evaluation at Enrollment and Termination.
  No Medical, Dental or Audiological adverse events.
Arm/Group | Medical, Dental, Audiological Safety 30 Days
Number analyzed (Participants) | 28
participants | 0

2. Primary Outcome: Efficacy: Ability to Understand Speech in Noise
Description: The primary efficacy outcome was a measure of the ability to understand speech in noise while wearing the device compared with not wearing the device. The Hearing in Noise Test (HINT) was utilized for this measure as it is the most widely used test for SSD devices. An improvement in HINT score is indicated as a negative (-) dB value change. A more negative (-dB) value indicates an improvement in understanding speech in noise. An improvement in a HINT score of -1 dB is equivalent to a 10% improvement in the ability to understand speech in noise and is likely of clinical benefit. The scores are calculated as HINT Advantage (aided compared with unaided) which depict the differences of using a device as compared to not wearing a device.
Time Frame: Day 1, Day 30
Measure: Mean (Standard Deviation); unit: dB
Groups:
- HINT (dB) Advantage: Effectiveness was defined as "Change from Baseline" analysis of the Hearing in Noise Test (HINT), Noise on Better Side Scores between without the BCD at day one and with the BCD at day thirty.Effectiveness was determined as an improvement in the HINT score for which the device was designed, that is, the condition where noise originates on the normal hearing side and speech is presented from the front. .
  An improvement in HINT score is indicated as a negative (-) dB value change. A change in the HINT score of -1 dB represents an improvement of 10% in speech intelligibility in that particular test condition. A 10% improvement in speech intelligibility in this very adverse listening condition is a noticeable benefit to the SSD subject. This amount of improvement is even more of a benefit in more realistic, less adverse listening conditions.
Arm/Group | HINT (dB) Advantage
Number analyzed (Participants) | 28
dB | -2.5 (1)
Statistical Analysis 1: Comparison: HINT (dB) Advantage; The endpoint was the calculated difference between the HINT result for the unaided condition prior to the 30-day trial period (Day 1) and the HINT result using the SoundBite (aided) at the end of the 30-day trial period (Day 30); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.5, Standard Deviation 1

3. Secondary Outcome: Measure of Benefit of SoundBite Using Abbreviated Profile of Hearing Aid Benefit (APHAB).
Description: The measure of the benefit of the device was assessed using the Abbreviated Profile of Hearing Aid Benefit (APHAB), a 24-item self-assessment inventory in which the amount of difficulty in everyday situations is reported with larger numbers indicating more difficulty. Device benefit is calculated by subtracting the score obtained after using a device from the score obtained before using the device. A software program is utilized to score the APHAB and results are compared a different time points. The APHAB is well characterized and broadly used as a quantifiable measurement of device benefit. The APHAB benefit scores can range from -99 (treatment worse than no treatment) to +99 (treatment better than no treatment)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Global Benefit Score
Groups:
- Global Benefit: The Global Benefit APHAB at 30 days is the change in APHAB scores between the unaided score at the start of the study and the APHAB score after 30 days of therapy. The APHAB questionnaire produces an overall Global score (GBL). The benefit provided by the SoundBite System can be determined by comparing changes in the mean APHAB score. The larger the APHAB benefit score the great the benefit. A negative APHAB score represents therapy resulting in a worse outcome than no therapy.
Arm/Group | Global Benefit
Number analyzed (Participants) | 28
Global Benefit Score | 18.80 (13.36)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Incidence of device- and procedure-related adverse events at 30 days
Groups:
- Incidence of Device- and Procedure-related Adverse Events: Incidence of device- and procedure-related adverse events at 30 days
Arm/Group | Incidence of Device- and Procedure-related Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days